CLINICAL TRIAL: NCT02552446
Title: Indirect Calorimetry an Essential Tool in the Intensive Care: Comparison of the Energy Expenditure Calculated With Different Body Weights Used in Several Predictive Equations and Indirect Calorimetry Measurements
Brief Title: Energy Expenditure in ICU Patients Using Predictive Formulas and Various Body Weights Versus Indirect Calorimetry
Status: Completed | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, HEIDEGGER CP, MD Deputy head physician, University Hospital, Geneva
Other Study IDs: CE:14-070; 13-18 (Other Grant/Funding Number: APSI)
Record Dates: First submitted 2015-08-25; First posted 2015-09-17 (Estimated); Last update posted 2015-09-17 (Estimated); Status verified 2015-09

CONDITIONS: Critical Illness; Body Weights
MeSH Terms: conditions — Critical Illness; Body Weight

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All patients: All ICU patients mechanically ventilated staying more than 72 hours were included and indirect calorimetry was performed and compared to predictive energy expenditure formulas using different body weights.

SUMMARY:
Indirect calorimetry is the gold standard to measure energy expenditure. In fact it is not always available and inconstantly feasible. Various equations for predicting energy expenditure based on body weights have been created. This study aims at determining the best suitable predictive strategy unless indirect calorimetry is available.

DETAILED DESCRIPTION:
Several clinical studies have shown that energy deficit as well as overfeeding lead to an increased risk of complications, especially infections, and increased mortality. The gold standard for determining energy expenditure in intensive care patients is indirect calorimetry. This method is expensive and requires a trained team for its use. In addition the reliability of the measurements depends on the clinical situation and may not be feasible (e.g. inspiratory O2 fraction >60%, end expiratory pressure > 9cmH2O, presence of bronchial gap, etc.). Moreover, there is no longer on the market valid indirect calorimeter for clinical use in mechanically ventilated patients, and the maintenance of the old valid one (Deltatrac II®) becomes increasingly problematic because the lack of spare parts. Intensivists have no more choice and use prediction equations for energy expenditure which are based on imprecise anthropometric data (height, weight). Especially for obese or malnourished patients in the intensive care the body weight represents not a reliable data. Similarly, secondary water inflation due to metabolic stress and resuscitation complicates the determination of the real body weight. The difficulty is to know which weight to use in predictive equations. Due to the paucity in literature on this subject, there is currently no consensus on the reference weight to use in the determination of nutritional needs and medication doses. So each prescriber calculates the energy target by taking a reference weight based on his own convictions. This study is part of a quality process of care and practices harmonization, aiming to identify the reference weight to be used and the best suited predictive equation, to predict energy expenditure for patients who cannot benefit from an indirect calorimetry.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the Geneva ICU
* Length of stay > 72 hours
* Mechanical ventilation with: FiO2 < 60%; positive end expiratory pressure < 9 cmH2O; no air leaks, absence of pulmonary multi-resistant bacteria
* Without mechanical ventilation: no claustrophobia; no oxygen dependence

Exclusion Criteria:

* All patients without inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICU ventilated patients of a tertiary mixed ICU population
Sampling Method: Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2014-04; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Best energy expenditure prediction, compared to indirect calorimetry by Deltatrac II vs. various predictive equations based on different body weights (ideal, anamnestic, actual, and adjusted). | Time frame will be 24 hours; no further follow-up will be done.
  Find the best energy expenditure prediction, by comparing results from an indirect calorimetry measurement using the Deltatrac II (considered the reference method), and various predictive equations based on body weight. The ideal body weights (calculated for a body mass index at 22.5 and 25 kg/m2, calculated with the Brocca and Lorentz equations and calculated with the Metropolitan Life Insurance tables), the anamnestic body weight (recorded from the patient/his family members or the electronical medical file), the actual body weight (using a built- in bed scale), and adjusted body weight (determined by correcting the measured body weight according to the cumulative fluid balance) will be recorded and used to calculate various predictive energy expenditure.

CONTACTS AND LOCATIONS:
Overall Officials: Claudia - Paula Heidegger, MD, Principal Investigator — University Hospital, Geneva
Locations (1):
- Service of Intensive Care, Geneva University Hospital,, Geneva, Switzerland

REFERENCES:
- [Derived] Graf S, Pichard C, Genton L, Oshima T, Heidegger CP. Energy expenditure in mechanically ventilated patients: The weight of body weight! Clin Nutr. 2017 Feb;36(1):224-228. doi: 10.1016/j.clnu.2015.11.007. Epub 2015 Nov 26. PMID 26653566